CLINICAL TRIAL: NCT01760109
Title: Phase IV Study on Piperacillin Sodium and Sulbactam Sodium for Injection(2:1) for Treatment of Respiratory and Urinary System Infection
Brief Title: Piperacillin Sodium and Sulbactam Sodium for Injection(2:1) for Treatment of Respiratory and Urinary System Infection
Acronym: PIP-SBT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiangbei Welman Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002HL0153
Record Dates: First submitted 2012-12-19; First posted 2013-01-03 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Tract Infections; Urinary Tract Infections
Keywords: Respiratory and urinary tract infections; Piperacillin Sodium and Sulbactam Sodium for Injection (2:1); Phase IV
MeSH Terms: conditions — Respiratory Tract Infections; Urinary Tract Infections | interventions — Piperacillin; Sulbactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Piperacillin Sodium and Sulbactam Sodium (Experimental): Drug:xintemie 1.5-3.0g,iv,bid 7-14 days
  serious infections 6.0-12.0g,iv,tid for 7-14 days
  Interventions: Drug: Piperacillin Sodium and Sulbactam Sodium

INTERVENTIONS:
Drug: Piperacillin Sodium and Sulbactam Sodium — 1.5-3.0g,iv,bid 7-14 days serious infections 6.0-12.0g,iv,tid for 7-14 days
  Other Names: xin te mie; te mie jun; xin ke jun

SUMMARY:
In the proposed study, the investigators plan to evaluate the efficacy and safety of Piperacillin Sodium and Sulbactam Sodium for Injection(2:1) for the treatment of respiratory and urinary tract acute bacterial infection.

DETAILED DESCRIPTION:
Piperacillin sodium and sulbactam sodium for injection (2:1)plays a therapeutic role by the former inhibiting bacterial cell wall synthesis，the latter making irreversible competitive inhibition of β-lactamase.The antimicrobial effect of Piperacillin can be enhanced by the two combined. The compound specifically aims to the mechanism of bacterial resistance, extending the life of Piperacillin in the treatment-resistant pathogen infections.

ELIGIBILITY:
Inclusion Criteria:

1. patients who qualify for moderate and severe acute respiratory or urinary tract bacterial infection of acute bacterial infections need for systemic antibiotic therapy.
2. Age>18 years old, Gender: both
3. Women of childbearing age were to be negative pregnancy test and agree to take contraceptive measures during the trial;
4. patients were volunteers and signed informed consent form;
5. patients did not participate in other clinical trials.

Exclusion Criteria:

1. Patients were hypersusceptibility to the test drug or other penicillins ,β-lactamase inhibitor
2. Pregnant and Lactating women
3. Patients have severe liver,kidney,cardiovascular,cerebrovascular,endocrine and hematopoietic system of primary diseases and that of immunodeficiency,advanced cancer or mental illness.
4. Patients who were complicated by other diseases and thought to affect efficacy evaluations or poor compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2011-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The rate of bacterial clearance | two years
  end of treatment of bacteriological efficacy(bactercial clearance) The fore-and-aft changes of clinical symptoms and signs after discontinuation of durgs

SECONDARY OUTCOMES:
Number of participants with Adverse Events | two years
  the incidence(%)of allergies, skin rashes, shock,death, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Changqing Li, doctor, Principal Investigator — Chongqing Red Cross Hospital
Locations (1):
- Chongqing Red Cross hospital, Chongqing, China